CLINICAL TRIAL: NCT01405157
Title: Phase 1, Open-label, Randomized, Single-dose, 2-treatment, Crossover Be Study Comparing Constituted Methylprednisolone Powder For Oral Suspension 4 Mg/ml To Methylprednisolone 16 Mg Tablet Under Fasting Conditions
Brief Title: A Bioequivalence Study Comparing Methylprednisolone Suspension To Methylprednisolone Tablets Under Fasting Conditions
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B0121007
Record Dates: First submitted 2011-07-25; First posted 2011-07-29 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Therapeutic Equivalency
Keywords: bioequivalence study; methylprednisolone; suspension; tablets; fasting
MeSH Terms: conditions — Fasting | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- methylprednisolone suspension (Experimental)
  Interventions: Drug: methylprednisolone
- methylprednisolone tablets (Active Comparator)
  Interventions: Drug: methylprednisolone

INTERVENTIONS:
Drug: methylprednisolone — constituted powder for oral suspension 4 mg/mL single dose at 16 mg
  Arms: methylprednisolone suspension
Drug: methylprednisolone — tablets 16 mg single dose
  Arms: methylprednisolone tablets

SUMMARY:
A study to determine whether a new formulation of methylprednisolone suspension is bioequivalent to methylprednisolone tablets under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between the ages of 21 and 55 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2 and a total body weight > 45 kg (99 lbs).

Exclusion Criteria:

* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive uring drug screen.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01-01 (Estimated); Primary Completion 2012-02-20 (Estimated); Study Completion 2012-02-20 (Estimated)

PRIMARY OUTCOMES:
AUCinf (area under the concentration time curve to infinity) | 0, 0.5, 1, 2, 3, 4, 5, 6, 10, 12, 16, 24 hours post dose
Cmax (maximum concentration) | 0, 0.5, 1, 2, 3, 4, 5, 6, 10, 12, 16, 24 hours post dose

SECONDARY OUTCOMES:
AUClast (area under the concentration time curve to last time point) | 0, 0.5, 1, 2, 3, 4, 5, 6, 10, 12, 16, 24 hours post dose
Tmax (time at maximum concentration) | 0, 0.5, 1, 2, 3, 4, 5, 6, 10, 12, 16, 24 hours post dose
Half-life | 0, 0.5, 1, 2, 3, 4, 5, 6, 10, 12, 16, 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0121007&StudyName=A%20Bioequivalence%20Study%20Comparing%20Methylprednisolone%20Suspension%20To%20Methylprednisolone%20Tablets%20Under%20Fasting%20Conditions%20